CLINICAL TRIAL: NCT07083206
Title: A Multi-center, Prospective, Non-intervention, Observational Study to Evaluate the Effectiveness and Safety of Switching to Pevarozet Tablet in Patients With Hypercholesterolemia Previously Treated With Atorvastatin or Rosuvastatin Monotherapy
Brief Title: A Study to Evaluate the Effectiveness and Safety of Fixed-Dose Combination of Pitavastatin/ Ezetimibe
Acronym: PIVOTAL
Status: Recruiting | Type: Observational
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Pitaeze_OS
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hypercholesterolemia; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of Pitavastatin/Ezetimibe FDC in patients with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Patients diagnosed with hypercholesterolemia who have been stably treated with atorvastatin or rosuvastatin monotherapy for at least 3 months, and for whom switching to fixed-dose combination pitavastatin/ezetimibe has been clinically decided
* Patients with available clinical laboratory test results related to efficacy and safety (TC, TG, HDL-C, LDL-C, AST, ALT, Cr/eGFR) within 12 months prior to switching to fixed-dose combination pitavastatin/ezetimibe (no changes in statin regimen or dosage during that period)
* Individuals (or their legally authorized representatives) who voluntarily provide written informed consent to participate in the study

Exclusion Criteria:

* Known hypersensitivity or history of hypersensitivity to any component of the investigational product
* Patients with active liver disease or persistent, unexplained elevations of aminotransferase levels
* Patients with severe hepatic impairment, biliary obstruction, or cholestasis
* Patients currently receiving cyclosporine treatment
* Patients diagnosed with myopathy
* Pregnant or breastfeeding women, or women who may be pregnant
* Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Any patient who, in the opinion of the investigator, is deemed unsuitable for study participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require administration of a fixed-dose combination of pitavastatin/ezetimibe for the treatment of hypercholesterolemia
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of reaching the target LDL-C level | 12 months after administration

CONTACTS AND LOCATIONS:
Overall Officials: Deok Kyu Cho, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) due to confidentiality concerns and lack of applicable data-sharing infrastructure.